CLINICAL TRIAL: NCT02457091
Title: Project GET FIT With MS: Guidelines for Exercise Training and Fitness Outcomes in MS
Acronym: GetFit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMSS IL-0010
Record Dates: First submitted 2014-03-17; First posted 2015-05-29 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; exercise; home-based; training; fitness
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Resistance Training; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stretching exercise (Active Comparator): The stretching condition will consist of 1-3 sets, 30-40 seconds of 12 stretching movements targeting lower body, upper body, and core areas performed 2 days per week.
  Interventions: Behavioral: Stretching exercise
- Resistance exercise (Experimental): The resistance condition will consist of 1-3 sets, 10-15 repetitions of 12 exercises targeting lower body, upper body, and core muscle groups performed 2 days per week.
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Behavioral: Resistance exercise — strength training consists of 1-3 sets , 10-15 repetitions of 10 exercises targeting lower body, upper body and core muscle groups
  Arms: Resistance exercise
Behavioral: Stretching exercise — The stretching condition will consist of 1-3 sets, 30-40 seconds of 12 stretching movements targeting lower body, upper body, and core areas performed 2 days per week.
  Arms: Stretching exercise

SUMMARY:
The purpose of this study is to test different types of exercise training for people with multiple sclerosis (MS). The exercise program is based on physical activity guidelines that have been developed specifically for people with MS. The investigators believe these guidelines will be effective for improving physical fitness and function in persons with mild-to-moderate MS.

DETAILED DESCRIPTION:
Most adults with multiple sclerosis (MS) are physically inactive. One approach to address physical inactivity in this population has involved the provision of physical activity guidelines. Such physical activity guidelines are an important tool for exercise prescription, promotion, and monitoring, and recommend that people with MS "participate in at least 30 minutes of moderate intensity aerobic activity 2 times per week and strength training exercises for major muscle groups 2 times per week." The guidelines were developed from a systematic literature review and have yet to be tested for efficacy in improving fitness or other outcomes. This study will test that efficacy of aerobic and resistance training alone and in combination (based on the MS physical activity guidelines) for improving physical fitness and other outcomes (e.g., walking, thinking, MS symptoms) in persons with MS who have mild-to-moderate disability. Such an examination will be important to confirm the efficacy of the exercise prescription for people with MS and health-care providers. The investigators will further perform an exploratory analysis of blood biomarkers and eye imaging parameters to examine some of the mechanisms of exercise training effects in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* a definite diagnosis of MS
* self-reported Expanded Disability Status Scale (EDSS) score < 6.0 or Patient Determined Disability Steps (PDDS) scale score ≤ 3.0
* relapse free in past 30 days
* willing and able to visit the University of Illinois at Urbana-Champaign for on seven occasions (two testing visits; five training visits) and participate in a 6-month home-based exercise program
* non-exerciser
* asymptomatic and physician approval for undertaking exercise testing and training

Exclusion Criteria:

* currently pregnant

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Physical fitness (aerobic and muscular) | 0 and 6 months
  Physical fitness determined by VO2 peak using a computer-driven cycle ergometer Muscular fitness determined by a seated dynamometer machine for leg strength and a hand dynamometer for upper body strength
Walking and physical function | 0 and 6 months
  A timed 25-Foot walk, a 6 -minute walk, walking on a GaitRite electronic walkway, 9-hole peg test and the use of a force platform will measure walking and physical function.
Cognition | 0 and 6 months
  The Brief International Cognitive Assessment for MS battery will be used.
Physical activity | 0 and 6 months
  an accelerometer along with the Godin Leisure Time Physical Activity Questionnaire and 7-day Physical Activity Recall Questionnaire will be used to measure physical activity.
Patient-rated outcomes | 0 and 6 months
  Self reporting questionnaires on fatigue, mobility, anxiety, depression, QoL, and social cognitive theory variable (e.g. Exercise Self-Efficacy Scale, Late-life function and disability scale)

SECONDARY OUTCOMES:
Body composition | 0 and 6 months
  DXA scan
OCT Eye imaging | 0 and 6 months
Cardiovascular function | 0 and 6 months
  ultrasonography techniques for arterial size, stiffness and blood pressure along with an ECG
Blood biomarkers | 0 and 6 months
  Circulating inflammatory markers, cytokines and growth factors

OTHER OUTCOMES:
Neurological examination | 0 and 6 months
Exercise training parameters | 24 weeks
  strength-training program or a stretching and limbering program

CONTACTS AND LOCATIONS:
Overall Officials: Lara Pilutti, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana-Champaign, Illinois, United States